CLINICAL TRIAL: NCT04240847
Title: Comparison of Skin Numbness and Kneeling Ability Between Midline Skin Incision Medial to Tibial Tubercle With Lateral to Tibial Tubercle Skin Incision in Simultaneous Bilateral Total Knee Arthroplasty
Brief Title: Comparison of Midline With Lateral Skin Incision in Simultaneous Bilateral TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Membership, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OrthoTU10
Record Dates: First submitted 2019-05-11; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Skin Numbness and Kneeling Ability
Keywords: skin incision; numbness; kneeling; total knee arthroplasty
MeSH Terms: conditions — Hypesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midline incision (Active Comparator): Skin incision at the midline, 1 cm medial to tibial tubercle
  Interventions: Procedure: Skin incision
- Lateral incision (Experimental): Skin incision at 1 cm lateral to tibial tubercle
  Interventions: Procedure: Skin incision

INTERVENTIONS:
Procedure: Skin incision — Skin incision on medial or lateral to tibial tubercle

SUMMARY:
This is a RCT which compare skin numbness, kneeling ability and functional outcome between midline incision and lateral incision in patients undergoing simultaneous bilateral TKA

ELIGIBILITY:
Inclusion Criteria:

* The patient undergoing simultaneous bilateral TKA
* Normal skin sensation on both knees
* Informed consent
* Good cognitive function

Exclusion Criteria:

* Previous surgical wound around the knee
* Peripheral vascular disease

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Skin numbness | 6 weeks, 3, 6 , 9, 12 months after surgery
  area of skin numbness
Kneeling ability | 6 weeks, 3, 6 , 9, 12 months after surgery
  Ability to kneel at 90 and 110 degrees on hard, firm and soft surface

SECONDARY OUTCOMES:
Functional outcome | 6 weeks, 3, 6 , 9, 12 months after surgery
  Modified WOMAC, Joint forgotten score
Knee range of motion | 6 weeks, 3, 6 , 9, 12 months after surgery
  flexion and extension angle of knee by goniometer
Incision length | 3 months
  Skin incision length at 90 degrees knee flexion
Complication | 6 weeks, 3, 6 , 9, 12 months after surgery
  chronic eczema at surgical wound

CONTACTS AND LOCATIONS:
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No